CLINICAL TRIAL: NCT07030491
Title: The Effect of Lactation Cookies on Breastfeeding Outcomes: A Pilot Randomized-Controlled Trial
Brief Title: The Effect of Lactation Cookies on Breastfeeding Outcomes in Lactating Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Notre Dame University - Louaize (Other)
Collaborators: Keserwan Medical Center (Other); Little Melly (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB 202425
Record Dates: First submitted 2025-05-29; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Breastfeeding
Keywords: Lactation; Breastfeeding; Galactagogues; Milk production; Randomized controlled trial; Lactation cookies
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups (lactation cookies or control cookies) and will remain in their group for the 30-day intervention period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactation Cookies (Experimental): Participants in this group will consume 2 lactation cookies daily for 30 days.
  Interventions: Other: Lactation Cookies
- Control Cookies (Placebo Comparator): Participants in this group will consume 2 control cookies (without active ingredients) daily for 30 days.
  Interventions: Other: Control Cookies

INTERVENTIONS:
Other: Lactation Cookies — Participants will consume 2 cookies per day (approximately 40g daily) for 30 consecutive days. The lactation cookies contain ingredients commonly believed to enhance milk production, including moringa, fenugreek, and ginger.
  Arms: Lactation Cookies
Other: Control Cookies — Participants in the control group will consume 2 cookies per day (approximately 40g total) for 30 consecutive days. These cookies are matched in taste, appearance, and caloric content but do not contain any known galactagogue ingredients.
  Arms: Control Cookies

SUMMARY:
The goal of this clinical trial is to learn if eating lactation cookies can help breastfeeding women make more milk. The main questions it aims to answer are:

* Do lactation cookies help increase milk production?
* Do lactation cookies make the breastfeeding experience easier or better?

Researchers will compare lactation cookies to regular cookies to see if lactation cookies work better.

Participants will:

* Eat 2 cookies every day for 30 days
* Visit the clinic 2 times, at the start and end of the study
* Keep a simple record of their breastfeeding and cookie eating

DETAILED DESCRIPTION:
Lactation cookies are popular among breastfeeding mothers because they often contain certain ingredients, such as fenugreek, ginger, and moringa, that are believed to help increase milk supply. Despite their widespread use, there is limited scientific evidence to confirm whether these cookies effectively increase breast milk volume or improve the breastfeeding experience.

This randomized controlled trial aims to evaluate the effects of lactation cookies on milk production and breastfeeding outcomes among exclusively breastfeeding mothers. Participants will be randomly assigned to consume a total of 2 cookies per day for 30 days; the cookies will either be lactation cookies or control cookies lacking milk-enhancing ingredients. Breast milk volume will be measured at the beginning and end of the study using standardized collection methods. Additional data will be collected to assess breastfeeding experience and any changes in infant feeding patterns.

This study will help clarify whether lactation cookies provide measurable benefits for breastfeeding mothers and their infants. The findings may support breastfeeding women and guide recommendations on the use of dietary galactagogues like lactation cookies.

ELIGIBILITY:
Inclusion Criteria:

* Women 1 month postpartum
* Exclusively breastfeeding
* Aged 18-45 years
* Healthy term infants (≥37 weeks gestation)
* Uncomplicated pregnancies and births
* Residing in Lebanon
* Planning to exclusively breastfeed for at least 2 months
* Intending to attend recommended pediatrician visits
* Infants must be at least 1 month old

Exclusion Criteria:

* Twin pregnancy
* Allergies or dislike of ingredients in the study cookies
* Presence of any health condition including: thyroid disease, epilepsy, psychosis, or bipolar disorder
* Currently receiving treatment for depression or anxiety
* Mastitis
* Smoking or alcohol consumption
* Taking medications or substances that may affect milk production, including: metoclopramide, chlorpromazine, domperidone, herbal galactagogues, thyroid hormones, or blood thinning medications

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological females
Enrollment: 36 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Change in breast milk volume from baseline to 1 month post-intervention | 1 month
  Breast milk volume will be assessed using the 3-hour milk expression protocol developed by Lai et al. (2010). This method involves hourly milk expression sessions over a 3-hour period, during which milk synthesis reaches a steady state, allowing for accurate estimation of the milk production rate.

SECONDARY OUTCOMES:
Change in breastfeeding self-efficacy scores from baseline to 1 month post-intervention | 1 month
  Assessed using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), a 14-item scale with scores ranging from 14 to 70, where higher scores indicate greater breastfeeding confidence.
Anxiety score changes from baseline to 1-month post intervention | 1 month
  Assessed using the State-Trait Anxiety Inventory (STAI), which includes two 20-item scales (State and Trait anxiety) scored 20-80; higher scores indicate higher anxiety levels.
Changes in perceived milk supply scores from baseline to 1-month post intervention | 1 month
  Assessed using the McCarter-Spaulding PIM questionnaire, with scores ranging from 5 to 50, where higher scores indicate greater perceived milk sufficiency.
Changes in postnatal depression scores from baseline to 1-month post intervention | 1 month
  Assessed using the Edinburgh Postnatal Depression Scale (EPDS), a 10-item scale with scores ranging from 0 to 30; higher scores indicate more severe depressive symptoms. Scores ≥13 suggest possible depression
Change in infant weight from baseline to 1 month post-intervention | 1 month
  Infant weight will be measured in kilograms (kg) using a calibrated infant scale by a pediatrician at baseline and after 1 month to assess changes in growth. Weight data will be interpreted using appropriate weight-for-age growth scores based on WHO growth standards.
Change in infant length from baseline to 1 month post-intervention | 1 month
  Infant length will be measured in centimeters (cm) using an infantometer or measuring board by a pediatrician at baseline and after 1 month to assess changes in linear growth. Length data will be interpreted using appropriate length-for-age growth scores based on WHO growth standards.
Change in infant head circumference from baseline to 1 month post-intervention | 1 month
  Infant head circumference will be measured in centimeters (cm) using a non-stretchable measuring tape by a pediatrician at baseline and after 1 month to assess brain growth and development. Head circumference data will be interpreted using appropriate head circumference-for-age growth scores based on WHO growth standards.
Change in number of wet diapers from baseline to 1 month | 1 month
  The number of wet diapers per day will be recorded by the mother using self-reported logs throughout the 1-month intervention period to assess hydration status and feeding adequacy.
Change in number of soiled diapers from baseline to 1 month | 1 month
  The number of soiled diapers per day will be recorded by the mother using self-reported logs throughout the 1-month intervention period to assess digestive health and feeding adequacy.
Change in breast milk composition from baseline to 1 month post-intervention | 1 month
  A 15 milliliter (mL) sample of breast milk will be collected from the mother at baseline and after 1 month to assess changes in milk composition. Analyses will focus on nutrient content and the potential transfer of bioactive components from the lactation cookies, including macronutrients (grams per liter, g/L), omega-3 fatty acids (milligrams per deciliter, mg/dL), and other relevant biomarkers.
Change in infant weight before and after each feed from baseline to 1 month post-intervention | 1 month
  Infant weight will be measured in kilograms (kg) using a calibrated infant scale immediately before and after each feeding session at baseline and later on Day 30. The difference between pre- and post-feed weights will be calculated to estimate milk intake per feed.

CONTACTS AND LOCATIONS:
Overall Officials: Jessy El Hayek, PhD, Principal Investigator — Notre Dame University
Locations (1):
- Keserwan Medical Center, Jounieh, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roznowski DM, Wagner EA, Riddle SW, Nommsen-Rivers LA. Validity of a 3-Hour Breast Milk Expression Protocol in Estimating Current Maternal Milk Production Capacity and Infant Breast Milk Intake in Exclusively Breastfeeding Dyads. Breastfeed Med. 2020 Oct;15(10):630-638. doi: 10.1089/bfm.2019.0182. Epub 2020 Jul 16. PMID 32700964
- [Background] Lai CT, Hale TW, Simmer K, Hartmann PE. Measuring milk synthesis in breastfeeding mothers. Breastfeed Med. 2010 Jun;5(3):103-7. doi: 10.1089/bfm.2009.0074. PMID 20433368
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] McCarter-Spaulding DE, Kearney MH. Parenting self-efficacy and perception of insufficient breast milk. J Obstet Gynecol Neonatal Nurs. 2001 Sep-Oct;30(5):515-22. doi: 10.1111/j.1552-6909.2001.tb01571.x. PMID 11572532
- [Background] Palacios AM, Cardel MI, Parker E, Dickinson S, Houin VR, Young B, Allison DB. Effectiveness of lactation cookies on human milk production rates: a randomized controlled trial. Am J Clin Nutr. 2023 May;117(5):1035-1042. doi: 10.1016/j.ajcnut.2023.03.010. Epub 2023 Mar 14. PMID 36921902